CLINICAL TRIAL: NCT06083272
Title: VitalThings Guardian Contactless Monitoring
Acronym: VINCENT
Status: Completed | Type: Observational
Sponsor: VitalThings (Industry)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 527859713
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Depression; Respiratory Failure; Deterioration, Clinical
Keywords: respiratory rate; patient monitoring; ultra wideband radar; contactless monitoring; medical device regulation
MeSH Terms: conditions — Respiratory Insufficiency; Clinical Deterioration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population: The study population is comprised of two subgroups;
  1. Adult patients admitted to the Emergency Ward (EW). Patients are recruited after the treatment and examination in EW are finished and the patient is waiting for transfer to a hospital ward.
  2. If there is a prolonged period of waiting time for a control blood sample, chest CT or any other examination which usually incurs significant waiting time in the EW. This will be evaluated by a specialist in emergency medicine based on the premise that the inclusion in the study will not delay or interfere with these examinations.
  Interventions: Device: Vitalthings Guardian M10 fixed and M10 mobile

INTERVENTIONS:
Device: Vitalthings Guardian M10 fixed and M10 mobile — VitalThings Guardian M10 / M10 mobile (VitalThings, Norway), are the investigational devices. These are the same technical devices made in two versions: one wall-mounted (VitalThings Guardian M10 fixed) and one mounted on a trolley (VitalThings Guardian M10 mobile). The Nox T3s and Nonin will be used as comparator devices.
  Other Names: Nox T3s (NOX Medical, Alpharetta, GA, USA ) with a Nonin 3150 pulse oximeter (Nonin Medical Inc., MN, USA)

SUMMARY:
This is a confirmatory study without any intervention. It is an uncontrolled, non-randomized and open-label study with measurements made with comparators, and it has a preset hypothesis for the primary endpoint. There are no similar devices to VitalThings Guardian M10 / M10 mobile on the market, consequently one or more different types of devices must be used as comparators.

DETAILED DESCRIPTION:
The purpose of the clinician investigation is to validate a claim made for the investigational device performance. The objective is to confirm that the device performs at +/- 1.2 respirations per minute (RPM) accuracy against the identified comparator device, and compare performance to the standard of care as documented in the literature. The study will be conducted with patients admitted to the emergency ward after the initial treatment and examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the Emergency Ward (EW)

Exclusion Criteria:

* Under age (below 18 years) and subjects not able to provide informed consent themselves. Subjects dismissed from the EW rooms within 30 minutes from first registration are removed from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The EW study population is beneficial to the study as it offers an unfiltered study population with a broad cross-section of potential admission reasons and diagnoses in a short period of time. Any patient that needs acute treatment/examination (typically triaged as "red") will per standard of care go into dedicated EW rooms and not be part of this study. The safe participation of each patient will be evaluated by a specialist in emergency medicine (PI) before invitation to participate.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Accuracy | Will be assessed after last participant has finished the investigation. One interim analysis in first week is planned.
  Documented system respiration frequency in RPM for both investigational device and comparator.

SECONDARY OUTCOMES:
Comparative pulse data | Will be assessed in 2024, furter details not established.
  Gather comparative pulse data to be used for retrospective validation of algorithm performance for contactless heart rate measurement/monitoring.

OTHER OUTCOMES:
Acceptance criteria respiratory rate | Will be assessed after last participant has finished the investigation. One interim analysis in first week is planned.
  A limit of agreement of ±1.2 RPM against comparators in setting the respiration rate.

CONTACTS AND LOCATIONS:
Overall Officials: Line Pedersen, MD, Phd, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toften S, Kjellstadli JT, Kvaerness J, Pedersen L, Laugsand LE, Thu OKF. Contactless and continuous monitoring of respiratory rate in a hospital ward: a clinical validation study. Front Physiol. 2024 Nov 27;15:1502413. doi: 10.3389/fphys.2024.1502413. eCollection 2024. PMID 39665054